CLINICAL TRIAL: NCT00261573
Title: The Safety and Efficacy of Galantamine in the Treatment of Vascular and Mixed Dementia
Brief Title: A Study of the Safety and Effectiveness of Galantamine Versus Placebo in the Treatment of Patients With Vascular Dementia or Mixed Dementia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006034
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-11

CONDITIONS: Alzheimer Disease; Vascular Dementia
Keywords: Alzheimer's disease with cerebrovascular disease ("mixed" dementia); probable vascular dementia; galantamine
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular; Mixed Dementias | interventions — Galantamine

INTERVENTIONS:
Drug: galantamine hydrobromide

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of galantamine (a drug for treating dementia) compared to placebo in the treatment of patients with dementia related to cerebrovascular disease (vascular dementia) or dementia related to Alzheimer's disease with cerebrovascular disease ("mixed" dementia).

DETAILED DESCRIPTION:
This multicenter, double-blind, placebo-controlled study will evaluate the safety and effectiveness of galantamine in patients with dementia related to cerebrovascular disease or related to Alzheimer's disease with cerebrovascular disease ("mixed" dementia). All patients will initially receive placebo for a 1-month period and then will receive galantamine (starting at a low dose and gradually increasing over 5 weeks to 12 mg twice daily) or placebo for 6 months. The primary measures of effectiveness include the change from baseline to the end of treatment in the ADAS-cog/11 score (Alzheimer's Disease Assessment Scale: sum of 11 cognitive items) and the CIBIC-plus score (Clinician's Interview Based Impression of Change - Plus Caregiver Input). Additional measures of effectiveness include the change from baseline to the end of the treatment in the ADAS-cog/13 score (Alzheimer's Disease Assessment Scale: sum of 13 cognitive items), the Disability Assessment for Dementia (DAD) score, and the Neuropsychiatric Inventory (NPI)) score. Safety evaluations (incidence of adverse events, electrocardiograms (ECGs), physical examinations, laboratory tests) will be performed throughout the study. Patients who complete the double-blind portion of the study will have the opportunity to participate in a 6-month open-label extension study in which they will receive galantamine for an additional 6 months. Effectiveness will be assessed after 6 weeks, 3 months and 6 months of open-label treatment. Safety evaluations (incidence of adverse events, ECGs, physical examinations, laboratory tests) will be performed throughout the open-label portion of the study. The study hypothesis is that galantamine will be effective in the treatment of patients with vascular or mixed dementia and will be well tolerated. Double-blind: Galantamine 12 mg or placebo by mouth twice daily for 6 months, starting at a low dose and gradually increasing over 5 weeks to the final dose; Open-label: galantamine 12 mg by mouth twice daily, starting at a low dose and gradually increasing over 6 weeks to the final dose.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of vascular dementia according to the NINDS-AIREN International Workshop criteria or with a diagnosis of "mixed" dementia (possible Alzheimer's disease with cerebrovascular disease) according to the NINCDS-ADRDA criteria
* mild-to-moderate dementia (score of 10 - 25 on the Mini Mental Status Exam (MMSE) and ADAS-cog score of at least 12)
* having the opportunity to perform activities of daily living (such as dressing, bathing, etc), including patients living independently in residential homes for the elderly
* had onset of disease between ages 40 - 90
* have a consistent informant to accompany them on scheduled visits

Exclusion Criteria:

* Neurogenerative disorders such as Parkinson's disease
* cognitive impairment resulting from conditions such as acute cerebral trauma, cerebral damage due to a lack of oxygen, vitamin deficiency, infections such as meningitis or AIDS, significant endocrine or metabolic disease, mental retardation, or a brain tumor
* having significant psychiatric disease, active peptic ulcer, clinically significant liver, kidney or lung disorders, or heart disease
* history of epilepsy, convulsions, drug abuse or alcohol abuse
* females of child bearing potential without adequate contraception

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 593 (Actual)
Dates: Start 1998-12; Study Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of double-blind treatment in ADAS-cog/11 (Alzheimer's Disease Assessment Scale: sum of 11 cognitive items) and CIBIC-plus (Clinician's Interview Based Impression of Change - Plus Caregiver Input) scores

SECONDARY OUTCOMES:
Change from baseline to the end of double-blind treatment in ADAS-cog/13, NPI, and DAD scores; Change in ADAS scores from baseline to end of open-label treatment; Incidence of adverse events; Changes in laboratory tests, ECGs and physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Erkinjuntti T, Kurz A, Gauthier S, Bullock R, Lilienfeld S, Damaraju CV. Efficacy of galantamine in probable vascular dementia and Alzheimer's disease combined with cerebrovascular disease: a randomised trial. Lancet. 2002 Apr 13;359(9314):1283-90. doi: 10.1016/S0140-6736(02)08267-3. PMID 11965273
- [Derived] Lim AWY, Schneider L, Loy C. Galantamine for dementia due to Alzheimer's disease and mild cognitive impairment. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD001747. doi: 10.1002/14651858.CD001747.pub4. PMID 39498781
- See also: A study of the safety and effectiveness of galantamine in patients with dementia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=702&filename=CR006034_CSR.pdf